CLINICAL TRIAL: NCT00490828
Title: Influence of Hydrocortisone on Humoral and Cellular Immunologic Markers in High Risk Patients After Cardiac Surgery
Brief Title: Influence of Hydrocortisone on Immunologic Markers and Health Care Related Quality of Life in Patients After Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Prof. Dr. Gustav Schelling, Ludwig-Maximilians University, Dept. of Anaesthesiology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 149/00
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2008-09

CONDITIONS: Systemic Inflammatory Response Syndrome; Posttraumatic Stress Disorder
Keywords: Cardiac surgery; systemic inflammatory response syndrome; health-related quality of life
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Stress Disorders, Post-Traumatic | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator)
  Interventions: Drug: Hydrocortisone
- B (Active Comparator): Stress doses of hydrocortisone
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone — Hydrocortisone
  Other Names: Stress doses of hydrocortisone

SUMMARY:
Hydrocortisone has been shown to improve the early outcome of high risk patients after cardiac surgery. A potential mechanism resulting in this effect may be its immunomodulatory action. In this prospective interventional study this hypothesis is to be proven.

DETAILED DESCRIPTION:
Methods: Prospective interventional randomized double blind placebo controlled study.

Intervention: Hydrocortisone in stress doses vs. placebo

Patients: 92 high risk patients after cardiac surgery

Measurements: Cytokines, Toll-like receptors, NF kappa B, outcome data, health care related quality of life, PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative left ventricular ejection fraction below 39 % duration of the extracorporeal circulation more than 97 min

Exclusion Criteria:

* Pregnancy
* Severe liver insufficiency
* Severe renal insufficiency
* Insulin dependent diabetes mellitus
* Steroid therapy
* Psychiatric disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-06; Primary Completion 2008-05 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
immunologic markers, health care related quality of life, PTSD | one and a half year

SECONDARY OUTCOMES:
early clinical outcome parameters (LOS in the ICU) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Shananz Azad, M.D., Principal Investigator — Department of Anesthesiology
Locations (1):
- Department of Anesthesiology, University of Munich, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Gibbison B, Villalobos Lizardi JC, Aviles Martinez KI, Fudulu DP, Medina Andrade MA, Perez-Gaxiola G, Schadenberg AW, Stoica SC, Lightman SL, Angelini GD, Reeves BC. Prophylactic corticosteroids for paediatric heart surgery with cardiopulmonary bypass. Cochrane Database Syst Rev. 2020 Oct 12;10(10):CD013101. doi: 10.1002/14651858.CD013101.pub2. PMID 33045104
- [Derived] Hauer D, Weis F, Campolongo P, Schopp M, Beiras-Fernandez A, Strewe C, Giehl M, Toth R, Kilger E, Schelling G. Glucocorticoid-endocannabinoid interaction in cardiac surgical patients: relationship to early cognitive dysfunction and late depression. Rev Neurosci. 2012;23(5-6):681-90. doi: 10.1515/revneuro-2012-0058. PMID 23006898